CLINICAL TRIAL: NCT03398031
Title: Magnesium Supplement in Early Pregnancy After ICSI
Brief Title: Effect of Magnesium Supplement in Early Pregnancy After ICSI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ashams university
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: ICSI
MeSH Terms: interventions — Magnesium Oxide; Magnesium; Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium supplement (Active Comparator): 90 female pregnant after ICSI after biochemical diagnosis of pregnancy will receive 500 mg magnesium supplement
  Interventions: Drug: Magnesium Oxide
- placebo (Placebo Comparator): 90 female pregnant after ICSI after biochemical diagnosis of pregnancy will receive placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Magnesium Oxide — After biochemical diagnosis of pregnancy each participant will receive magnesium plus 500 mg tablet once daily till the end of the 1st trimester
  Other Names: magnesium plus tablet
  Arms: Magnesium supplement
Drug: Placebo Oral Tablet — After biochemical diagnosis of pregnancy each participant will receive placebo tablet once daily till the end of the 1st trimester
  Arms: placebo

SUMMARY:
Daily supplement of magnesium after biochemical diagnosis of pregnancy in females pregnant after ICSI and through out 1st trimester

DETAILED DESCRIPTION:
a fall of magnesium levels at 2-3 weeks of gestation. This drop of magnesium concentration is larger following IVF as compared to spontaneous pregnancies.

so magnesium supplement start after biochemical diagnosis of pregnancy and throughout the 1st trimester

ELIGIBILITY:
Inclusion Criteria:

* age 25_38 years
* BMI 25_30

  * females pregnant after ICSI after biochemical diagnosis of pregnancy

Exclusion Criteria:

* females with poor ovarian reserve and poor responders

  * abnormality in uterine cavity detected by hysteroscopic evaluation pre ICSI and not treated
  * hydrosalpinx

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
1st trimesteric abortion | 13 week of gestation
  Either spontaneous or missed abortion

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt

IPD SHARING:
Plan to Share IPD: No